CLINICAL TRIAL: NCT00642161
Title: A Placebo-controlled Comparison of the Efficacy, Safety and Pharmacokinetics of the Current US Version of Pulmicort (Budesonide) Turbuhaler and the New Version of Pulmicort Turbuhaler in Asthmatic Children and Adolescents.
Brief Title: New Version Pulmicort Turbuhaler USA Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-004-0726; D5254C00726
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort; Children; Paediatrics; budesonide; Flexhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: budesonide
  Other Names: Pulmicort

SUMMARY:
A comparison of the safety, efficacy and budesonide pharmacokinetics of the currently approved Pulmicort Turbuhaler with a new version of the inhaler, in children and adolescents who have asthma. In addition the study evaluated the functionality of the new inhaler at the end of its intended life.

ELIGIBILITY:
Inclusion Criteria:

* Male or females aged 6 to 17 with a diagnosis of asthma for at least 3 months. Have used inhaled corticosteroids for no more than one month before entering the study or none at all.
* A forced expiratory volume (FEV1) in 1 second of 75% to 90% of predicted normal for those aged 6 to 11 and 60% to 90% for those aged 12 to 17 years.
* Airway reversibility of at least 12% , use of orally inhaled corticosteroids for no more than one month immediately before entering the study or none at all.

Exclusion Criteria:

* Life threatening asthma, Two or more overnight hospitalisations for asthma within 1 year or any emergency room visit for asthma within 6 months of starting study.
* Use of steroid tablets or injections during the month prior to Visit 1 and use of other asthma medicines (except rescue medication) within 2 weeks prior to the study.
* Any acute exacerbation of asthma or a respiratory tract infection within 30 days prior to Visit 1. Must not smoke or have smoked.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Estimated)
Dates: Start 2002-11; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in % predicted Forced Expiratory Volume in 1 second | Week 2, 4 and 8, then at week 12

SECONDARY OUTCOMES:
Change from baseline in Forced Vital Capacity, Morning Peak Expiratory Flow, Daytime and nighttime asthma symptom scores, beta-agonist use and discontinuation rate | Week 2, 4 and 8, then at week 12
Incidence of Adverse Events | Week 2, 4 and 8, then at week 12
Pharmacokinetics of budesonide (AUC, maximum concentration and time to maximum concentration | 6 or 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Andersson, Study Director — AstraZeneca employee; Lars-Göran Carlsson, Study Director — AstraZeneca employee